CLINICAL TRIAL: NCT05253690
Title: Comparing Two Methods for Inserting a Balloon Catheter : View-guided Approach Using a Speculum Versus Manual Guided Approach at Cervical Examination - a Prospective Randomized Trail
Brief Title: Comparing Methods for Balloon Catheter Inserting: View Guided (Speculum) Versus Manual Guided at Cervical Examination
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Principal Investigator, Dr. Maya Wolf, Director of fetal maternal unit, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0150-21-NHR
Record Dates: First submitted 2022-01-19; First posted 2022-02-24 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Cervical Ripening
Keywords: labor induction; balloon catheter; cervical ripenning; speculum
MeSH Terms: interventions — Labor, Induced

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Who Masked: Outcomes Assessor
Masking Description: The obstetrician evaluating labor progress is blinded for type of intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- speculum guided (Active Comparator): view-guided approach using a speculum
  Interventions: Procedure: balloon catheter insertion approach for labor induction
- manual guided (Experimental): manual guided approach at cervical examination
  Interventions: Procedure: balloon catheter insertion approach for labor induction

INTERVENTIONS:
Procedure: balloon catheter insertion approach for labor induction — Parous women will be randomized to labor induction by view-guided approach using a speculum for catheter insersion versus manual guided catheter balloon insersion at cervical examination

SUMMARY:
Induction of labor is a common obstetric procedure. Foley catheter is recommended by WHO for cervical ripening. Insertion is typically speculum guided but digital insertion has been reported to be faster, better tolerated and with similar insertion success rate compared to speculum guided insertion in a mixed population of nulliparas and multiparas. We evaluated the ease, maternal satisfaction and success rate of digital compared to speculum guided insertion of Foley catheter for induction of labor in parous women with unripe cervixes based on Bishop score<6.

DETAILED DESCRIPTION:
Globally, there has been an increase in birth-induced labor from 9.5% to 29% in the last 3 decades. Circumstances requiring induction include gestational age of 41 weeks or more, hypertension, fetal growth disorder, gestational diabetes and others.

There are different methods of induction, the choice of the best method depends on the bishop score, an estimate based on cervical related data like opening (cm), deletion (%) and other parameters, also the choice of induction method depends on the obstetric history of the mother. Bishop score less than 6, indicates an immature cervix, and therefore increases the chance of induction failure.

The mechanism by which the catheter works includes a mechanical effect that causes the cervix to dilate, but in addition the direct stress on the inner surface of the cervix tissue and lower segment of the uterus indirectly causes local secretion of prostoglandins which help softening the cervix and may induce contractions.

Inserting a single or double balloon catheter, is traditionally performed in a lithotomy position, and after inserting a speculum, disinfecting with polydine, identifying the external os of the cervix and then inserting the catheter, inflating the balloon with saline up to 30-80 ml while looking at the position of the balloon.

Insertion of the catheter is typically speculum guided, but digital insertion has been reported to be faster, better tolerated and with similar insertion success and infections rate compared to speculum guided insertion in a mixed population of nulliparas and multiparas. We evaluate the ease, maternal satisfaction and success rate of digital compared to speculum guided insertion of Foley catheter for induction of labor in parous women with unripe cervixes based on Bishop score<6.

Methods: A randomized trial. Participants are parous at term with unripe cervixes (Bishop Score ≤ 6) admitted for induction of labor. They will be randomized to digital or speculum-aided transcervical Foley catheter insertion in lithotomy position (1:1, 50 in each group). Primary outcomes are pain score [VAS] and time to birth. Secondary outcomes are procedure duration, maternal satisfaction, success and bishop score change.

ELIGIBILITY:
Inclusion Criteria:

Singelton parous women Term pregnancy Vertex position

-

Exclusion Criteria:

Nulliparous women previous cesarean section Prom twins pregnancy Fetal anomaly

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Enrollment: 100 (Estimated)
Dates: Start 2022-01-10 (Actual); Primary Completion 2025-01-10 (Estimated); Study Completion 2025-01-10 (Estimated)

PRIMARY OUTCOMES:
Maternal pain sensation during the procedure | during the procedure
  VAS (visual analog scale) SCORE scale 0-10 0-better outcome 10-worse outcome
induction to delivery duration | through study completion, an average of 1 year
  hours

SECONDARY OUTCOMES:
catheter insertion duration | during the procedure
  minutes
maternal satisfaction- questionnaire | during one hour after the procedure
  questionnaire including 5 questions about maternal preference for catheter insertion methods
chorioamnionitis- fever during labor | during labor up to 48 hours
  clinical diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Maya Wolf, MD, Study Director — Galilee Medical Center
Locations (1):
- Galil Medical Center, Nahariya, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jonsson M, Hellgren C, Wiberg-Itzel E, Akerud H. Assessment of pain in women randomly allocated to speculum or digital insertion of the Foley catheter for induction of labor. Acta Obstet Gynecol Scand. 2011 Sep;90(9):997-1004. doi: 10.1111/j.1600-0412.2011.01197.x. Epub 2011 Jun 27. PMID 21615714
- [Background] Kuhlmann MJ, Spencer N, Garcia-Jasso C, Singh P, Abdelwahab M, Vaughn M, Marshall K, Prasad N, Soulsby-Monroy R, Saade GR, Saad AF. Foley Bulb Insertion by Blind Placement Compared With Direct Visualization: A Randomized Controlled Trial. Obstet Gynecol. 2021 Jan 1;137(1):139-145. doi: 10.1097/AOG.0000000000004182. PMID 33278290
- [Background] Chia HM, Tan PC, Tan SP, Hamdan M, Omar SZ. Speculum versus digital insertion of Foley catheter for induction of labor in Nulliparas with unripe cervix: a randomized controlled trial. BMC Pregnancy Childbirth. 2020 May 29;20(1):330. doi: 10.1186/s12884-020-03029-0. PMID 32471369
- [Background] Liu X, Wang Y, Zhang F, Zhong X, Ou R, Luo X, Qi H. Double- versus single-balloon catheters for labour induction and cervical ripening: a meta-analysis. BMC Pregnancy Childbirth. 2019 Oct 16;19(1):358. doi: 10.1186/s12884-019-2491-4. PMID 31619189
- [Background] de Vaan MD, Ten Eikelder ML, Jozwiak M, Palmer KR, Davies-Tuck M, Bloemenkamp KW, Mol BWJ, Boulvain M. Mechanical methods for induction of labour. Cochrane Database Syst Rev. 2019 Oct 18;10(10):CD001233. doi: 10.1002/14651858.CD001233.pub3. PMID 31623014
- [Derived] Abu Shqara R, Nakhleh Francis Y, Haj H, Markdorf S, Lowenstein L, Frank Wolf M. Digital vs speculum-guided catheter balloon insertion for cervical ripening in multiparas: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Jun;5(6):100943. doi: 10.1016/j.ajogmf.2023.100943. Epub 2023 Mar 25. PMID 36972835